CLINICAL TRIAL: NCT07167069
Title: Comparison of Treatment Adherence and Toxicities of HIV Positive Patients Versus HIV Negative Cervical Cancer Patients in India
Brief Title: India HIV-CervCa Project
Status: Active, not recruiting | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Tata Memorial Hospital (Other Government); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: UPCC 20824; 834664 (Other: The University of Pennsylvania Institutional Review Board); DAA3-19-65331-1 (Other: National Institute of Allergy and Infectious Diseases (NIAID))
Record Dates: First submitted 2025-08-19; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: HIV Positive; HIV Negative; Cervical Cancer
Keywords: Chemotherapy; Concurrent Chemoradiotherapy; Radiotherapy
MeSH Terms: conditions — HIV Seropositivity; Uterine Cervical Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy specimens collected for Tumor-Infiltrating Lymphocytes (TILs) detection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV Positive: Cervical Cancer Patients with HIV positive
  Interventions: Radiation: Radiation Therapy
- HIV Negative: Cervical Cancer Patients with HIV negative
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Standard of Care Chemoradiation for Cervical cancer patients in India.

SUMMARY:
The investigators propose to prospectively study the difference in treatment (CTRT) completion and toxicities between HIV positive and HIV negative women in India with locally advanced cervical cancer receiving CTRT.

DETAILED DESCRIPTION:
This study will compare chemoradiation completion rates for cervical cancer in two groups, women with HIV and women without HIV. The investigators will also be analyzing tumor tissue for tumor infiltrating lymphocytes which are thought to be involved in disease progression.

ELIGIBILITY:
Inclusion Criteria:

* patients with newly biopsy proven squamous carcinoma or adenocarcinoma of the uterine cervix, FIGO stage IB2-IIIB in whom curative CTRT is planned
* Karnofsky performance status ≥ 70
* Patients with lower paraortic lymph nodes (below the level of L2 vertebra)
* patients diagnosed with cervical cancer whom also HIV positive or HIV negative

Exclusion Criteria:

* patients with active tuberculosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cervical cancer at Tata Memorial Hospital in India.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Completion Rates of Cancer Treatment | 2 years
  To evaluate and compare the completion rates of cancer treatment in HIV positive cervical cancer patients and HIV negative cervical cancer patients.
  Treatment adherence is defined as receiving at least 5 cycles of weekly cisplatin chemotherapy and completion of all prescribed radiation (including brachytherapy) and chemotherapy within 8 weeks of treatment initiation.
Impact of HIV Infection on acute toxicities | 2 years
  To compare the incidence of acute grade ≥3 gastrointestinal, genitourinary and hematological toxicities using CTCAE v4 in patients receiving concurrent cisplatin-based chemo-radiation and brachytherapy for cervical cancer in HIV positive and HIV negative patients. Acute toxicities include any toxicity occurring within 90 days of treatment completion.

SECONDARY OUTCOMES:
Tumor infiltrating lymphocytes (TILs) | 2 Years
  To identify and characterize tumor infiltrating lymphocytes (TILs) with reference to numbers and phenotype in tumor biopsies of HIV positive and HIV negative cervical cancer patients in India

CONTACTS AND LOCATIONS:
Overall Officials: Surbhi Grover, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No